CLINICAL TRIAL: NCT02665572
Title: Outcome of Renal Transplant on a Defunctionalized Bladder. A Randomized Controlled Trial
Brief Title: Outcome of Renal Transplant on a Defunctionalized Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Zahran, Assistant lecturer of urology and renal transplantation, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zahran MH3182015
Record Dates: First submitted 2015-10-29; First posted 2016-01-28 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Renal Transplantation Into a Defunctionalized Bladder
Keywords: renal transplantation; defunctionalized bladder; bladder recycling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- renal transplant without bladder recycling (No Intervention): the patients allocated to this arm and met inclusion criteria will undergo renal transplant without prior recycling of the bladder
- renal transplantation with bladder recycling (Active Comparator): the patients allocated in this arm will undergo bladder recycling prior to renal transplantation
  Interventions: Behavioral: bladder recycling

INTERVENTIONS:
Behavioral: bladder recycling — Bladder recycling will be done by the patient after proper education. It will be started by the instillation of the sterile water in the bladder in amount equal to the estimated bladder capacity. Then the amount will be gradually increased till the patient can withstand filling the bladder with 300 cc of sterile water for 2 hours.
  Arms: renal transplantation with bladder recycling

SUMMARY:
In this study, investigators will prospectively evaluate the outcome of renal transplantation into a defunctionalized bladder by comparing direct transplantation into this defunctionalized bladder and pre-transplant programmed bladder cycling.

DETAILED DESCRIPTION:
Study population:

The study will include patients maintained on hemodialysis for more than 12 months, have oliguria or anuria, reduced bladder capacity, have no history of lower urinary tract dysfunction and have no evidence of urological cause of renal failure. Patients with history of lower urinary tract symptoms before developing renal failure and those with lower urinary tract disease resulting in renal failure will be excluded.

Study design:

It is a randomized controlled trial comparing the outcome of programmed bladder cycling before the time of renal transplantation and direct transplantation without bladder cycling in patients with defunctionalized bladder. Patients, who meet the inclusion criteria, will be randomly allocated into two groups. The first group will undergo renal transplantation on the defunctionalized bladder without bladder recycling. The second group will undergo renal transplantation after bladder recycling.

Measurements:

All patients will be diagnosed by proper history taking, cystoscopy, ascending cystogram and cystometry in order to confirm the diagnosis of reduced bladder capacity and exclude any organic or neurological cause. Bladder recycling will be done by the patient after proper education. It will be started by the instillation of the sterile water in the bladder in amount equal to the estimated bladder capacity. Then the amount will be gradually increased till the patient can withstand filling the bladder with 300 cc of sterile water for 2 hours. Any associated complications will be reported and the time needed to reach the due bladder capacity will be recorded. The procedure of renal transplantation will be carried out according to the hospital protocol and the ureteroneocystostomy will be done by a non-stented Leich Gregoir technique.

Assuming that the bladder will regain its activity and full capacity after 8 weeks of transplantation, all patients will be assessed 3 months after transplantation by the following:

1. IPSS questionnaire in order to evaluate the lower urinary tract symptoms.
2. Ascending cystogram.
3. Cystometry.
4. Graft function.

Outcome:

The primary outcome is to evaluate whether bladder recycling is efficient to restore bladder function prior to renal transplantation in terms of IPSS score, and urodynamic evaluation. The secondary outcome is to evaluate the differences in graft and patients outcome between groups.

Power calculation and Statistical analysis:

We hypothesized that at 3 months postoperatively; recipients without bladder training will be non-inferior to those underwent bladder training in terms of cystometric capacity. Based on this, to achieve a difference in mean cystometric capacity of 50 cc in favor of bladder training patients, 16 patients in each group are required to achieve a power of 80% and an α error of 0.05. Statistical power is determined using medcalc version 12.5.0.0 software and all statistical analyses will be performed using IBM version 20 statistical software.

ELIGIBILITY:
Inclusion Criteria:

* patients maintained on hemodialysis for more than 12 months
* have oliguria or anuria
* reduced bladder capacity
* have no history of lower urinary tract dysfunction and have no evidence of urological cause of renal failure.

Exclusion Criteria:

* Patients with history of lower urinary tract symptoms before developing renal failure and
* those with lower urinary tract disease resulting in renal failure will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-08; Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
improvement of bladder function after recycling | 3 months
  to evaluate whether bladder recycling is efficient to restore bladder function prior to renal transplantation by urodynamic evaluation and ascending cystogram to measure the bladder capacity in cm

SECONDARY OUTCOMES:
voiding function after renal transplantation | 3 months after renal transplantation
  1. IPSS questionnaire in order to evaluate the lower urinary tract symptoms score ( score range from 0-35)
  2. Ascending cystogram.( capacity in cm, presence of reflux, postvoiding residual urine)
  3. Cystometry ( capacity in cm)
graft function | 1 year
  creatinine clearance and estimated GFR by renography ( ml/min/1.73 m2)

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Dakahlia Governorate, Egypt